CLINICAL TRIAL: NCT00838435
Title: A Phase 3b Open-Label Study to Evaluate the Effect of Kuvan® on Neurocognitive Function, Maintenance of Blood Phenylalanine Concentrations, Safety, and Population Pharmacokinetics in Young Children With Phenylketonuria
Brief Title: Effect of Kuvan on Neurocognitive Function, Blood Phenylalanine Level, Safety, and Pharmacokinetics in Children With PKU
Acronym: PKU-015
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-015
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Phenylketonuria
Keywords: Phenylketonuria; PKU; Kuvan; Phenoptin; Biopten; Neurocognitive Function; Phenylalanine
MeSH Terms: conditions — Phenylketonurias | interventions — sapropterin; phenoptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sapropterin dihydrochloride (Experimental): A dose of 20 mg/kg will be administered dissolved in water or apple juice, based on subject's age and ability, and taken orally once daily with food.
  Interventions: Drug: sapropterin dihydrochloride

INTERVENTIONS:
Drug: sapropterin dihydrochloride — A dose of 20 mg/kg will be administered dissolved in water or apple juice, based on subject's age and ability, and taken orally once daily with food.
  Other Names: Kuvan; Phenoptin; BH4; 6R BH4

SUMMARY:
This multicenter, open label study is designed to evaluate the safety of Kuvan® and its effect on neurocognitive function, blood Phe concentration, and growth in children with PKU who are 0-6 years old.

DETAILED DESCRIPTION:
Rigorous control of diet is typically advocated in children 4 years and under with PKU because brain sensitivity to high Phe concentrations is expected to be greatest during these years of rapid neurocognitive development.

Prolonged high blood Phe concentrations are neurotoxic and lead to impairment of intelligence and other brain functions (such as attentiveness). Reduction of blood Phe concentrations through dietary control is an important determinant of long-term neurologic outcome in PKU patients, and reduction of blood Phe concentrations in patients with PKU has been shown to decrease the long term risk of neurologic injury.

It is difficult for many patients to maintain reduced blood Phe, and many patients with PKU experience some degree of neurological impairment despite efforts to maintain dietary Phe control.

The strongest determinant of intelligence quotient (IQ) and cognitive function is compliance with blood Phe control. Several clinical studies with Kuvan have already demonstrated efficacy in reducing blood Phe in subjects older than 4 years. This study will examine whether addition of Kuvan to the standard of care at an early age in children with well controlled diets can lower blood Phe levels (ie, reach and maintain a goal of ≤ 240 micromole/L) and preserve neurocognitive functioning. In addition, this study will provide data on Kuvan exposure, rate of uptake, half life, and clearance in young children.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of PKU with hyperphenylalaninemia (HPA) documented in the medical record by at least 2 blood Phe concentrations greater than or equal to 360 micromole/L (6 mg/dL) taken at least 3 days apart
* Documented blood Phe control (defined by the standard used at each treatment center) prior to study enrollment, if applicable (eg, the subject is old enough for these data to be collected); blood Phe concentrations for subjects < 6 months old at Screening must be considered controlled and stable by the Investigator
* Willing to adhere to a prescribed Phe restricted diet in order to maintain blood Phe concentrations within the recommended ranges established at the subject's study site
* Age 0 to 6 years old, inclusive, at Screening
* Parent(s) or guardian(s) willing and able to provide written, signed informed consent after the nature of the study has been explained, and prior to any research-related procedures
* Parent(s) or guardian(s) willing and able to comply with all study procedures
* Female subjects of childbearing potential (as determined by the investigator) and sexually mature male subjects willing to use a medically accepted method of contraception throughout the study. Female subjects of childbearing potential willing to undergo periodic pregnancy tests during the course of the study

Exclusion Criteria:

* Established diagnosis of primary tetrahydrobiopterin (BH4) deficiency
* Known hypersensitivity to Kuvan or its excipients
* History of organ transplantation
* Perceived to be unreliable or unavailable for study participation or to have parents or legal guardians who are perceived to be unreliable or unavailable
* Use of methotrexate or other medications that inhibit folate metabolism
* Serious neuropsychiatric illness (eg, major depression) not currently under medical control
* Use of Kuvan or any investigational agent within 30 days prior to Screening, or known requirement for any investigational agent prior to completion of all scheduled study assessments
* Concurrent disease or condition that would interfere with study participation or safety (eg, seizure disorder, oral steroid-dependent asthma or other condition requiring oral or parenteral corticosteroid administration, or insulin dependent diabetes)
* Any condition that, in the view of the Principal Investigator (PI), renders the subject at high risk for failure to comply with treatment or to complete the study
* Use of phosphodiesterase type 5 (PDE5) inhibitor.

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2009-02; Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lilienstein, M.D., Study Director — BioMarin Pharmaceutical
Locations (19):
- United States (12):
  - La Jolla, California
  - Orange, California
  - Tampa, Florida
  - Chicago, Illinois
  - Boston, Massachusetts
  - Kansas City, Missouri
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Nashville, Tennessee
  - Salt Lake City, Utah
  - Milwaukee, Wisconsin
- Canada (7):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted at 20 sites in the U.S. and Canada.
Groups:
- Sapropterin Dihydrochloride: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
  Part 1: 95 subjects participated in Part 1.
  Pharmacokinetic (PK) Sub-Study: 94 subjects participated in the PK substudy, one subject declined participation.
  6-month Safety/Efficacy Sub-Study: 65 subjects met the minimum required score of 80, Kuvan responders, all 65 subjects participated in Safety/Efficacy Substudy.
  Part 2: 65 subjects met the minimum required score of 80 at baseline (Month 2) neurocognitive tests, all 65 subjects participated in Part 2.
Period: Part 1 (4 Weeks)
Arm/Group | Sapropterin Dihydrochloride
Started | 95
Completed | 95
Not Completed | 0
Period: PK Sub-Study 2 (4 Weeks)
Arm/Group | Sapropterin Dihydrochloride
Started | 94 (1 subject declined participation in the PK Sub-Study.)
Completed (of the 95 who started Part 1.) | 93
Not Completed | 1
Not completed — no postdose blood sample | 1
Period: Safety/Efficacy Sub-Study 1 (6 Months)
Arm/Group | Sapropterin Dihydrochloride
Started | 65 (65 of 95 subjects in Part 1 were determined responders & eligible for the Safety/Efficacy Sub-study.)
Completed | 63
Not Completed | 2
Not completed — Adverse Event | 2
Period: Part 2 (7 Years)
Arm/Group | Sapropterin Dihydrochloride
Started | 65 (65 of 95 subjects in Part 1 were determined responders & eligible for the Part 2 of the study.)
Completed | 49
Not Completed | 16
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 1
Not completed — Sponsor Decision | 6
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Population: Safety Population consist of all subjects who received any study drug in the Full Analysis Set(FAS).
Groups:
- Sapropterin Dihydrochloride: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.2 (1.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 89
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Black or African American | 2
  White | 79
  Other | 9
Weight [Mean (Standard Deviation); unit: kg] | 15.6 (6.08)
Height [Mean (Standard Deviation); unit: cm] | 94.8 (17.70)

OUTCOME MEASURES:

1. Primary Outcome: Full-Scale Intelligence Quotient (FSIQ) Score
Description: Full Scale Intelligence Quotient (FSIQ) is a score derived through administration of selected subtests from age appropriate Wechsler Intelligence assessments. Weschler Preschool and Primary Scale of Intelligence (WPPSI)-III is used for children >30 months and ≤6 years; and Weschler Intelligence Scale for Children (WISC)-IV is used for children >6 years old. The outcome variable will be the FSIQ score from WPPSI-III and/or WISC-IV tests.
  FSIQ results can range from 40 being the lowest and 160 being the highest. Higher scores are associated with higher intelligence quotient.
Time Frame: Assessments through 84 months.
Population: Efficacy population is based on all subjects from the enrolled population who have at least 2 WPPSI/ WISC assessments.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Kuvan 20 mg/kg Once Daily: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
  Part 2 (7 years): Part 1 determined that 71 subjects were Kuvan responders, defined as a 30% average reduction in blood Phe concentration during the first 4 weeks .This included 8 subjects who had Phe reductions less than 30% but were granted exemptions to participate in Part 2 of the study.
  Sixty-five of these 71 subjects were enrolled in Part 2. All 65 subjects met the minimum required FSIQ test score of ≥80 at baseline (Month 2).
Arm/Group | Kuvan 20 mg/kg Once Daily
Number analyzed (Participants) | 63
score on a scale
  FSIQ Baseline | 101.06 (14.039)
  FSIQ Month 12: number analyzed (Participants) | 59
  FSIQ Month 12 | 103.64 (13.202)
  FSIQ Month 24: number analyzed (Participants) | 58
  FSIQ Month 24 | 104.69 (11.697)
  FSIQ Month 36: number analyzed (Participants) | 55
  FSIQ Month 36 | 103.78 (12.759)
  FSIQ Month 48: number analyzed (Participants) | 48
  FSIQ Month 48 | 104.25 (13.242)
  FSIQ Month 60: number analyzed (Participants) | 38
  FSIQ Month 60 | 100.76 (14.280)
  FSIQ Month 72: number analyzed (Participants) | 23
  FSIQ Month 72 | 104.57 (11.012)
  FSIQ Month 84: number analyzed (Participants) | 27
  FSIQ Month 84 | 104.22 (12.236)
Statistical Analysis 1: Comparison: Kuvan 20 mg/kg Once Daily; A random coefficient model was used to calculate the slope (per year) of FSIQ over the entire study period. Factors in the model included visit and testing sequence, with change in FSIQ score as the dependent variable. Random terms include both intercept and visit. The treatment was considered successful if the lower 95% confidence limit of the mean change excluded a decline of greater than 5 points over a 2-year window; Test type: Other — Coefficient estimates from a random coefficient model and associated p-values; Slope = -0.5768, 95% CI 2-sided [-1.6004 to 0.4468] — The slope shown above is based on a 2-year window

2. Secondary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Adverse Event is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, and that does not necessarily have a causal relationship with this treatment.
  Drug Related Adverse all noxious and unintended responses to a medical product related to any dose. This means that a causal relationship between a medicinal product and an AE is at least a reasonable possibility, ie, the relationship cannot be ruled out.
  A serious adverse event (SAE) is an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect.
Time Frame: Up to 7 years
Population: Enrolled Population consists of all subjects who enter Part 2. This population involves subjects who respond to Kuvan and had a Bayley-III or IQ test score ≥80 within 6 weeks of determination of Kuvan responsiveness in Part 1. Kuvan 20 mg/kg once daily.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
  Part 2 (7 years): Sixty-five of the 71 subjects that were determined to be Kuvan responders in Part 1 were enrolled in Part 2. All 65 subjects met the minimum required IQ test score of ≥80 at baseline (Month 2).
Arm/Group | Part 2
Number analyzed (Participants) | 65
Participants
  Any Adverse Events (AEs) | 65
  Drug-Related Adverse Events | 35
  Any Serious Adverse Events | 11
  Drug-Related Serious Adverse Events | 2
  Any AEs causing study discontinuation | 2
  Drug-related AEs causing study discontinuation | 2
  Death | 0

3. Secondary Outcome: Change From Baseline in Growth Measurements - Height Z-Scores
Description: Z-scores of Height determined using World Health Organization(WHO) growth charts for children <24 months and Centers for Disease Control and Prevention(CDC) clinical growth charts for children 24 months and older.
  A height z-score is a standardized height measure after considering important factors like age and gender, in which higher z-scores are associated with taller children. Z-scores (or standard deviation scores) describe how far a measurement is from the median (mean). A z-score of 0 is the same as a 50th percentile; a positive value is a factor of standard deviation (SD) unit above the 50%; and a negative value is a factor of SD unit below 50%.
Time Frame: Baseline and up to 84 months
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Z-score change from baseline
Groups:
- Sapropterin Dihydrochloride: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
  Part 2 (7 years): Sixty-five of the 71 subjects that were determined to be Kuvan responders in Part 1 were enrolled in Part 2. All 65 subjects met the minimum required IQ test score of ≥80 at baseline (Month 2).
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 63
Z-score change from baseline
  Baseline | 0.4 (0.97)
  Change from Baseline Week 4: number analyzed (Participants) | 62
  Change from Baseline Week 4 | 0.0 (0.44)
  Change from Baseline Month 3: number analyzed (Participants) | 61
  Change from Baseline Month 3 | 0.1 (0.57)
  Change from Baseline Month 6: number analyzed (Participants) | 59
  Change from Baseline Month 6 | 0.1 (0.72)
  Change from Baseline Month 12: number analyzed (Participants) | 62
  Change from Baseline Month 12 | -0.1 (0.73)
  Change from Baseline Month 18: number analyzed (Participants) | 62
  Change from Baseline Month 18 | 0.0 (0.78)
  Change from Baseline Month 24: number analyzed (Participants) | 62
  Change from Baseline Month 24 | 0.0 (0.71)
  Change from Baseline Month 30: number analyzed (Participants) | 62
  Change from Baseline Month 30 | -0.1 (0.72)
  Change from Baseline Month 36: number analyzed (Participants) | 62
  Change from Baseline Month 36 | -0.1 (0.71)
  Change from Baseline Month 42: number analyzed (Participants) | 61
  Change from Baseline Month 42 | -0.1 (0.73)
  Change from Baseline Month 48: number analyzed (Participants) | 62
  Change from Baseline Month 48 | -0.2 (0.77)
  Change from Baseline Month 54: number analyzed (Participants) | 62
  Change from Baseline Month 54 | -0.2 (0.78)
  Change from Baseline Month 60: number analyzed (Participants) | 62
  Change from Baseline Month 60 | -0.2 (0.75)
  Change from Baseline Month 66: number analyzed (Participants) | 62
  Change from Baseline Month 66 | -0.2 (0.77)
  Change from Baseline Month 72: number analyzed (Participants) | 59
  Change from Baseline Month 72 | -0.3 (0.78)
  Change from Baseline Month 78: number analyzed (Participants) | 55
  Change from Baseline Month 78 | -0.2 (0.78)
  Change from Baseline Month 84: number analyzed (Participants) | 50
  Change from Baseline Month 84 | -0.2 (0.83)

4. Secondary Outcome: Change From Baseline in Growth Measurements - Weight Z-Scores
Description: Z-scores of Weight determined using World Health Organization(WHO) growth charts for children <24 months and Centers for Disease Control and Prevention(CDC) clinical growth charts for children 24 months or older.
  A weight z-score is a standardized weight measure after considering important factors like age and gender, in which higher z-scores are associated with heavier children. Z-scores (or standard deviation scores) describe how far a measurement is from the median (mean). A z-score of 0 is the same as a 50th percentile; a positive value is a factor of SD unit above the 50%; and a negative value is a factor of SD unit below 50%.
Time Frame: Baseline and up to 84 months
Population: Efficacy Population
Measure: Mean (Standard Deviation); unit: Z-score change from baseline
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 63
Z-score change from baseline
  Baseline | 0.4 (0.84)
  Change from Baseline Week 4 | 0.0 (0.24)
  Change from Baseline Month 3: number analyzed (Participants) | 55
  Change from Baseline Month 3 | 0.0 (0.26)
  Change from Baseline Month 6: number analyzed (Participants) | 61
  Change from Baseline Month 6 | 0.0 (0.36)
  Change from Baseline Month 12 | 0.1 (0.45)
  Change from Baseline Month 18: number analyzed (Participants) | 62
  Change from Baseline Month 18 | 0.1 (0.59)
  Change from Baseline Month 24: number analyzed (Participants) | 62
  Change from Baseline Month 24 | 0.1 (0.62)
  Change from Baseline Month 30: number analyzed (Participants) | 62
  Change from Baseline Month 30 | 0.1 (0.68)
  Change from Baseline Month 36: number analyzed (Participants) | 62
  Change from Baseline Month 36 | 0.1 (0.71)
  Change from Baseline Month 42: number analyzed (Participants) | 62
  Change from Baseline Month 42 | 0.0 (0.75)
  Change from Baseline Month 48: number analyzed (Participants) | 62
  Change from Baseline Month 48 | 0.0 (0.79)
  Change from Baseline Month 54: number analyzed (Participants) | 62
  Change from Baseline Month 54 | 0.0 (0.84)
  Change from Baseline Month 60: number analyzed (Participants) | 62
  Change from Baseline Month 60 | 0.0 (0.91)
  Change from Baseline Month 66: number analyzed (Participants) | 62
  Change from Baseline Month 66 | 0.0 (0.85)
  Change from Baseline Month 72: number analyzed (Participants) | 59
  Change from Baseline Month 72 | 0.0 (0.77)
  Change from Baseline Month 78: number analyzed (Participants) | 56
  Change from Baseline Month 78 | 0.0 (0.81)
  Change from Baseline Month 84: number analyzed (Participants) | 50
  Change from Baseline Month 84 | 0.0 (0.85)

5. Secondary Outcome: Change From Baseline in Growth Measurements - Head Circumference Z-Scores
Description: Z-scores of Head Circumference determined using World Health Organization(WHO) growth charts for children <24 months and Centers for Disease Control and Prevention(CDC) clinical growth charts for children 24 months and older.
  A head circumference z-score is a standardized head circumference measure after considering important factors like age and gender, in which higher z-scores are associated with children with larger heads. Z-scores (or standard deviation scores) describe how far a measurement is from the median (mean). A z-score of 0 is the same as a 50th percentile; a positive value is a factor of SD unit above the 50%; and a negative value is a factor of SD unit below 50%.
Time Frame: Baseline and up to 84 months
Population: Efficacy Population, subjects less than 36 months of age.
Measure: Mean (Standard Deviation); unit: Z-score change from baseline
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 33
Z-score change from baseline
  Baseline: number analyzed (Participants) | 31
  Baseline | 0.2 (0.95)
  Change from Baseline Week 4: number analyzed (Participants) | 29
  Change from Baseline Week 4 | 0.1 (0.69)
  Change from Baseline Month 3: number analyzed (Participants) | 26
  Change from Baseline Month 3 | 0.0 (0.40)
  Change from Baseline Month 6: number analyzed (Participants) | 28
  Change from Baseline Month 6 | 0.1 (0.70)
  Change from Baseline Month 12: number analyzed (Participants) | 22
  Change from Baseline Month 12 | 0.1 (0.56)
  Change from Baseline Month 18: number analyzed (Participants) | 15
  Change from Baseline Month 18 | -0.1 (1.00)
  Change from Baseline Month 24: number analyzed (Participants) | 10
  Change from Baseline Month 24 | 0.2 (0.74)
  Change from Baseline Month 30: number analyzed (Participants) | 6
  Change from Baseline Month 30 | 0.8 (0.81)

6. Secondary Outcome: Change From Baseline in Bayley-III Scores - Neurocognitive Testing Results
Description: The Bayley-III is a tool for assessing all facets of development in infants within an age range of 12 to 30 months, with normative data available for infants as young as 16 days. Composite scores are derived for cognitive, language, and motor development and scaled to a metric, with a range of 40 to 160. Higher scores are a better outcome.
Time Frame: At Month 6, 12, 18 and 24
Population: Efficacy Population, analysis only comprised of subjects less than 30 months of age.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 26
score on a scale
  Cognitive: Baseline | 102.31 (9.081)
  Cognitive: Change from Baseline Month 6: number analyzed (Participants) | 22
  Cognitive: Change from Baseline Month 6 | 5.68 (10.943)
  Cognitive: Change from Baseline Month 12: number analyzed (Participants) | 19
  Cognitive: Change from Baseline Month 12 | 2.11 (13.157)
  Cognitive: Change from Baseline Month 18: number analyzed (Participants) | 11
  Cognitive: Change from Baseline Month 18 | 2.27 (20.170)
  Cognitive: Change from Baseline Month 24: number analyzed (Participants) | 6
  Cognitive: Change from Baseline Month 24 | 0.83 (23.962)
  Language: Baseline | 100.73 (12.914)
  Language: Change from Baseline Month 6: number analyzed (Participants) | 22
  Language: Change from Baseline Month 6 | 2.59 (10.966)
  Language: Change from BaselineMonth 12: number analyzed (Participants) | 19
  Language: Change from BaselineMonth 12 | 1.37 (14.469)
  Language: Change from Baseline Month 18: number analyzed (Participants) | 11
  Language: Change from Baseline Month 18 | 4.82 (22.903)
  Language: Change from Baseline Month 24: number analyzed (Participants) | 6
  Language: Change from Baseline Month 24 | -3.00 (18.407)
  Motor: Baseline | 104.96 (11.837)
  Motor: Change from Baseline Month 6: number analyzed (Participants) | 22
  Motor: Change from Baseline Month 6 | 1.32 (10.952)
  Motor: Change from Baseline Month 12: number analyzed (Participants) | 19
  Motor: Change from Baseline Month 12 | 2.11 (12.297)
  Motor: Change from Baseline Month 18: number analyzed (Participants) | 11
  Motor: Change from Baseline Month 18 | 0.18 (19.894)
  Motor: Change from Baseline Month 24: number analyzed (Participants) | 6
  Motor: Change from Baseline Month 24 | 7.50 (18.512)

7. Secondary Outcome: Baseline Concentration of Tetrahydrobiopterin (BH4)(C0)
Description: Baseline concentration of BH4(C0) with associated inter-individual variability.
Time Frame: At predose and postdose - 0.22, 3.2 and 7 hours
Population: Eighty patients were evaluable from PKU-015 PK Sub-Study.
Measure: Least Squares Mean (Standard Error); unit: µg/L
Groups:
- Sapropterin Dihydrochloride: A dose of 20 mg/kg dissolved in water or apple juice, administered once daily orally, with food.
  Substudy 2 (Pharmacokinetics Substudy): 94 subjects participated in the PK substudy, one subject declined participation.
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 80
µg/L | 16.6 (4.1)

8. Secondary Outcome: Absorption Rate Constant (Ka) of Kuvan
Description: Population pharmacokinetic parameter, Absorption Rate Constant (Ka)
Time Frame: At predose and postdose - 0.22, 3.2 and 7 hours
Population: Eighty subjects were evaluable from PKU-015 PK Sub-Study.
Measure: Least Squares Mean (Standard Error); unit: l/hour
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 80
l/hour | 0.235 (23.8)

9. Secondary Outcome: Apparent Volume of Distribution (V/F) of Kuvan
Description: Population pharmacokinetic parameter apparent volume of distribution (V/F)
Time Frame: At predose and postdose - 0.22, 3.2 and 7 hours
Population: Eighty subjects were evaluable from PKU-015 PK Sub-Study.
Measure: Mean (Standard Error); unit: L
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 80
L | 1209 (56.4)

10. Secondary Outcome: Apparent Clearance (CL/F) of Kuvan
Description: Population pharmacokinetic parameter apparent clearance (CL/F)
Time Frame: At predose and postdose - 0.22, 3.2 and 7 hours
Population: Eighty subjects were evaluable from PKU-015 PK Sub-Study.
Measure: Mean (Standard Error); unit: L/hour
Arm/Group | Sapropterin Dihydrochloride
Number analyzed (Participants) | 80
L/hour | 815 (50.9)

ADVERSE EVENTS:
Time Frame: Up to 7 years
Groups:
- Safety Population: All subjects who enrolled in the study (Full Analysis Set) and received any study drug.
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 12/95
Other Adverse Events (participants affected / at risk) | 90/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=95)
Phenylketonuria (Congenital, familial and genetic disorders) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Croup infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 1
Airway complication of anaesthesia (Injury, poisoning and procedural complications) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Convulsion (Nervous system disorders) | 2
Autism spectrum disorder (Psychiatric disorders) | 1
Diet noncompliance (Social circumstances) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=95)
Lymphadenopathy (Blood and lymphatic system disorders) | 13
Ear pain (Ear and labyrinth disorders) | 7
Conjunctivitis (Eye disorders) | 9
Myopia (Eye disorders) | 5
Abdominal discomfort (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 17
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 39
Nausea (Gastrointestinal disorders) | 5
Teething (Gastrointestinal disorders) | 5
Toothache (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 53
Pain (General disorders) | 6
Pyrexia (General disorders) | 56
Seasonal allergy (Immune system disorders) | 11
Bronchitis (Infections and infestations) | 11
Conjunctivitis infective (Infections and infestations) | 7
Croup infectious (Infections and infestations) | 9
Ear infection (Infections and infestations) | 26
Gastroenteritis (Infections and infestations) | 28
Gastroenteritis viral (Infections and infestations) | 11
Hand-foot-and-mouth disease (Infections and infestations) | 7
Influenza (Infections and infestations) | 20
Lower respiratory tract infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 42
Otitis media (Infections and infestations) | 22
Pharyngitis (Infections and infestations) | 8
Pharyngitis streptococcal (Infections and infestations) | 19
Pneumonia (Infections and infestations) | 6
Rhinitis (Infections and infestations) | 6
Sinusitis (Infections and infestations) | 13
Streptococcal infection (Infections and infestations) | 7
Upper respiratory tract infection (Infections and infestations) | 55
Urinary tract infection (Infections and infestations) | 6
Viral infection (Infections and infestations) | 18
Fall (Injury, poisoning and procedural complications) | 6
Laceration (Injury, poisoning and procedural complications) | 7
Ligament sprain (Injury, poisoning and procedural complications) | 5
Procedural pain (Injury, poisoning and procedural complications) | 5
Red blood cell sedimentation rate increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Headache (Nervous system disorders) | 25
Anxiety (Psychiatric disorders) | 6
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 43
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 30
Dry skin (Skin and subcutaneous tissue disorders) | 6
Eczema (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 15
Urticaria (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2010-11-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT00838435/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT00838435/SAP_001.pdf